CLINICAL TRIAL: NCT02377375
Title: Deep Brain Stimulation (DBS) for Obsessive Compulsive Disorder (OCD) in the Bed Nucleus of the Stria Terminalis (BNST): Improving Targeting Precision
Brief Title: Deep Brain Stimulation (DBS) for Obsessive Compulsive Disorder (OCD): Improving Targeting Precision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S57471
Record Dates: First submitted 2015-01-27; First posted 2015-03-03 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micro-assisted (Experimental): In each patient, one electrode will be implanted using the standard technique and one electrode will be implanted using the micro-electrode assisted technique. The side is randomized.
  Interventions: Procedure: Micro-assisted technique
- Standard (Active Comparator): In each patient, one electrode will be implanted using the standard technique and one electrode will be implanted using the micro-electrode assisted technique. The side is randomized.
  Interventions: Procedure: Standard technique

INTERVENTIONS:
Procedure: Micro-assisted technique — Medtronic DBS lead 3391-28cm Medtronic electrode array microrecording 22670
  Arms: Micro-assisted
Procedure: Standard technique — Medtronic DBS lead 3391-28cm
  Arms: Standard

SUMMARY:
When comparing targeting precision between DBS in parkinsonian patients and OCD patients, an unexpected deviation from the planned targets was discovered in OCD patients (Nuttin et al., 2013). The objective of this trial is to investigate whether the use of a micro-electrode assisted technique improves targeting precision in DBS at the BNST.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OCD following the diagnostic and statistical manual of mental disorders-fourth edition (DSM-IV) criteria for OCD (300.3).
* Failure of documented trials of pharmacotherapy, following an appropriate treatment algorithm for OCD.
* Failure of documented trial of cognitive and behavioural therapy
* Duration of illness: min. 5 year
* Y-BOCS (Yale-Brown Obsessive Compulsive Scale) at least 30/40.
* Age: 20-65 year

Exclusion Criteria:

* DSM-IV diagnosis on axis 2 of severe personality disorder in cluster A or B, especially in the case of heightened risk for acting-out behavior.
* DSM-IV diagnosis on axis 3 of organic brain pathology or significant abnormalities on MRI.
* Present or past history of psychotic symptoms.
* Present substance abuse, or instable remission of substance abuses (i.e. no substance abuse during the last 12 months).
* Any disorder affecting cognitive functioning, other than motor tics and Gilles de la Tourette's Syndrome
* Mental retardation. A minimum threshold of cognitive skills is needed for adequate reporting on questionnaires and evaluation, and for technical handling of the instruments in a later faze.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Millimeter difference in position between planned and actual target | 4 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bart Nuttin, MD, PHD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Nuttin B, Gielen F, van Kuyck K, Wu H, Luyten L, Welkenhuysen M, Brionne TC, Gabriels L. Targeting bed nucleus of the stria terminalis for severe obsessive-compulsive disorder: more unexpected lead placement in obsessive-compulsive disorder than in surgery for movement disorders. World Neurosurg. 2013 Sep-Oct;80(3-4):S30.e11-6. doi: 10.1016/j.wneu.2012.12.029. Epub 2012 Dec 23. PMID 23268197